CLINICAL TRIAL: NCT04071912
Title: Isokinetic Muscular Assessment After ACL Ligamentoplasty: Study of Factors Predictive of Muscle Imbalance.
Acronym: PREDICT-ACL
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM U1075 COMETE, UNICAEN, Caen France (Unknown)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Chief Resident PM&R and Sport departments MD, MSc, University Hospital, Caen
Other Study IDs: PREDICT-ACL
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: ACL - Anterior Cruciate Ligament Deficiency; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL: All sports patients who had a muscle evaluation at 3-4 months and 6-8 months after ACL ligamentoplasty since January 2016

SUMMARY:
Despite advances in surgery and rehabilitation, the return to sport after anterior cruciate ligament (ACL) reconstruction surgery remains a major challenge.

challenge. Among the objective criteria retained, the isokinetic muscle strength assessment is an increasingly practiced evaluation and it is recommended to carry out follow-ups at 3-4 months (intermediate) and at 6-8 months (final) after surgery. However, the factors associated with muscle imbalance are uncertain and the threshold values of the intermediate isokinetic strength test (3-4 months) are inconsistent. In a retrospective analysis, the investigators aim to assess the predictive criteria for muscle imbalance after ACL reconstruction surgery.

DETAILED DESCRIPTION:
The investigators aim to retrospectively studied all sports patients who had a muscle evaluation at 3-4 months and 6-8 months after anterior cruciate ligament (ACL) reconstruction surgery since January 2016. The objective criterion were based on the international guidelines for muscle imbalance after ACL surgery and return to sport, as a muscle deficit of less than 20% on knee extensor muslces and less than 10% on knee flexor muscles of the operated knee (vs. healthy).

The investigators will study the predictive analysis of the intermediate muscle strength test to predict the risk of muscle imbalance on the final isokinetic muscle strength assessment. The investigators will also study the individual, injury and surgical criteria associated with muscle imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an ACL reconstruction surgery (isolated or associated with other meniscal or ligamentary surgery)
* Patient included in the sport medicine follow-up protocole with intermediate and final isokinetic muscular assessment at 3-4 months and 6-8 mnths after surgery respectively
* Patient who received the information form

Exclusion Criteria:

* Patient who did not participate in all follow-up consultations and isokinetic muscular assessments
* Cognitive or sensory impairment making it impossible to understand the information form
* Neurological, traumatic or osteoarticular history responsible for muscle imbalance prior to surgery

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All sports patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 3-4 months and 6-8 months after ACL reconstruction surgery since January 2016
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Strength | ACL group: Two evaluations on both injured and healthy knees: (1) 3 months after surgery and (2) 7 months after surgery; Routine practice following guidelines
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.

SECONDARY OUTCOMES:
Individual characteristics | ACL group: Two follow-up medical consultations: (1) 3 months after surgery and (2) 7 months after surgery; Routine practice following guidelines
  Personal characteristics recorded in the medical report as age, gender, type of sport and sport level of practice and return to sport after the surgery
Injury characteristics | ACL group: Two follow-up medical consultations: (1) 3 months after surgery and (2) 7 months after surgery; Routine practice following guidelines
  Injury characteristics recorded in the medical report as the type of injury (ACL only, ACL and meniscus, ACL with other ligament injury, recurrent ACL injury) the time before surgery, the type of rehabilitation before and after surgery
Surgery characteristics | ACL group: Two follow-up medical consultations: (1) 3 months after surgery and (2) 7 months after surgery; Routine practice following guidelines
  Surgery characteristics recorded in the medical report as the type of surgery, the surgery duration and tourniquet time

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drigny J, Ferrandez C, Gauthier A, Guermont H, Praz C, Reboursiere E, Hulet C. Knee strength symmetry at 4 months is associated with criteria and rates of return to sport after anterior cruciate ligament reconstruction. Ann Phys Rehabil Med. 2022 Jun;65(4):101646. doi: 10.1016/j.rehab.2022.101646. Epub 2022 Apr 30. PMID 35167984